CLINICAL TRIAL: NCT07053176
Title: Usefullnes of Local Lidocaine Paravertebral Cervical Injection on Cervicogenic Dizziness Symptoms Management: a Randomzied Clinical Trial
Brief Title: Impact of Local Lidocaine Paravertebral Cervical Injection on Cervicogenic Dizziness Symptoms
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Uniter Onlus (Other)
Responsible Party: Principal Investigator, Alessandro Micarelli, UNITER ONLUS, Uniter Onlus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NeuralCGD1
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Cervicogenic Dizziness
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): patients will received lidocaine paravertebral injection
  Interventions: Drug: 0.5% Lidocaine
- Sham (Placebo Comparator): patients will received saline solution paravertebral injection
  Interventions: Drug: Saline Solution (NaCl 0,9%)

INTERVENTIONS:
Drug: 0.5% Lidocaine — 0.5% lidocaine injection will be administered in the paravertebral intramuscular region with 12 mm, 30 G needle from C2 to C7 bilaterally
  Arms: Lidocaine
Drug: Saline Solution (NaCl 0,9%) — saline solution will be administered bilaterally in the paravertebral intamuscular region from C2 to C7 with 12 mm 30 G needle
  Arms: Sham

SUMMARY:
at least 42 patients affected by cervicogenic dizziness will be allocated to the experimental group or in the placebo group. in the first group patients will received 2 paravertebral intramuscular injection of lidocaine 0.5% while in the placebo group they will received saline solution with the same injection technique. patients will be evaluated by subjective and objective testing before the treatment, immediatly and 3 months after the treatment.

DETAILED DESCRIPTION:
at least 42 patients affected by cervicogenic dizziness will be allocated to the experimental group or in the placebo group. in the first group patients will received 2 paravertebral intramuscular injection of lidocaine 0.5% while in the placebo group they will received saline solution with the same injection technique. patients will be evaluated by subjective and objective testing before the treatment, immediatly and 3 months after the treatment. subjective testing will include dizziness handicap inventory, Neck Disability Index, Neck Pain Intensity, Tampa Scale for Kinesiophobia, Hospital Anxiety and Depression Scale. Objective testing will include cervical range of motion, joint position error and static posturography testing.

ELIGIBILITY:
Inclusion Criteria:

1) presence of a subjective feeling of dizziness associated with pain, movement, rigidity, or certain positions of the neck at least from 3months; 2) Cervical pain, trauma, and/or disease (3) If from traumatic origin, there has to be a temporal proximity between the onset of dizziness and the neck injury.

Exclusion Criteria:

1. Exclusion of these differential diagnoses: (a) Migrainous vertigo (b) Vertigo of central origin (c) Benign paroxysmal positional vertigo (d) Meniere disease (e) Vestibular neuritis (f) Vertigo induced by drugs (g) Psychogenic vertigo (anxiety and/or panic disorder and/or phobia) (h) Orthostatic hypotension
2. presence of trauma or recent surgery in the head, face, neck, or chest; an otorhinolaryngological diagnosis of central or peripheral vertigo, and receiving physiotherapy or other treatment during the study period.
3. allergy to lidocaine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | one monthe
  Dizziness Handicap Inventory version comprises 25 questions designed to assess a patient's functional (9 questions), emotional (9 questions), and physical (7 questions) limitations on a three-point scale, with higher scores reflecting greater perceived handicap

SECONDARY OUTCOMES:
Neck Disability Index | one month
  This is conceived in a single-factor structure including 10 items to survey different activities of daily living on a 6-point Likert-type scale (from 0 to 5). Higher values score more severe pain and worse disability.
Neck Pain Intensity | one month
  Neck Pain Intensity will be assessed by means of the visual analogue scale for pain. This reliable tool is conceived as a 100-mm horizontal line between the extremes 'no pain' and 'worst imaginable pain', on the left and on the right respectively.
Tampa Scale for Kinesiophobia | one month
  Within this 17 item self-report tool each question will be scored using a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree); 4 questions (4, 8, 12 and 16) were negatively worded and reversely scored. Higher values score a higher degree of kinesiophobia.
Hospital Anxiety and Depression Scale. | one month
  This self-administered tool includes 14 questions, rated on a 4-point Likert type scale (from 0 to 3 points), with higher scores reflecting abnormal anxiety and depression levels. The questionnaire encompasses two subscales of seven items that evaluate anxiety and depression, respectively
The 36-item short form survey (SF-36) | one month
  The 36-item short form survey (SF-36) was used for general health-related quality of life (Qol) assessment. the sf-36 is an established, validated, generic instrument that measures health-related Qol in diverse patient populations. it is based on a 36-item questionnaire with eight subscales and two component summaries of physical and mental health related QOL.
Cervical range of motion | one month
  A cervical range of motion goniometer (Performance Attainment Associates, 3550 Lahore Rd, St Paul, MN), which has been shown to be a reliable tool with good validity, will be used to measure cervical spine movements. Active flexion, extension, left and right rotation, and left and right lateral flexion have been measured three times and then averaged
Static posturography testing | one month
  Each patient will be instructed to keep an upright position on a standardized platform for static posturography (ED800 Medi-Care Solutions S.R.L. Euroclinic). The recording period will be 60s for each test (eyes closed or open while standing on the stiff platform) and the sampling frequency in the time domain was 25Hz. The center of pressure will be monitored, while performing the test. The posturographic parameters considered in our study will be the trace length (length), the surface of the ellipse of confi dence (surface),
Cervical relocation test (CRT) | one month
  This test will be used to evaluate cervical proprioception. According to previous protocols, a headlamp with an integrated laser pointer is placed in the centre of the patient's forehead. The subject keeps a neutral head and neck position as he seats at 90cm from a wall in front of him. The point emitted by the laser pointer is then centred on a target fixed on the wall. We will use the target created by Rob Landel. With his eyes closed, the subject turns his head to the right, comes back to the initial position, and indicates verbally when he thinks his head is centred. Left rotation, flexion, and extension were also evaluated. Each movement is repeated three times and the patient opens his eyes and re-centers on the target between each measure. To assess the patient's result, we will calculated the mean distance in centimetres between eachpoint and the centre of the target, for each head position.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniter Onlus, Fara in Sabina, Rieti, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Micarelli A, Viziano A, Carlino P, Granito I, Micarelli RX, Alessandrini M. Reciprocal roles of joint position error, visual dependency and subjective perception in cervicogenic dizziness. Somatosens Mot Res. 2020 Dec;37(4):262-270. doi: 10.1080/08990220.2020.1803257. Epub 2020 Aug 10. PMID 32772608
- [Background] Karadas O, Inan LE, Ulas U, Odabasi Z. Efficacy of local lidocaine application on anxiety and depression and its curative effect on patients with chronic tension-type headache. Eur Neurol. 2013;70(1-2):95-101. doi: 10.1159/000350619. Epub 2013 Jul 2. PMID 23839118
- [Background] Raeissadat SA, Rayegani SM, Sadeghi F, Rahimi-Dehgolan S. Comparison of ozone and lidocaine injection efficacy vs dry needling in myofascial pain syndrome patients. J Pain Res. 2018 Jun 29;11:1273-1279. doi: 10.2147/JPR.S164629. eCollection 2018. PMID 29988746
- [Background] Mellick LB, Mellick GA. Treatment of acute orofacial pain with lower cervical intramuscular bupivacaine injections: a 1-year retrospective review of 114 patients. J Orofac Pain. 2008 Winter;22(1):57-64. PMID 18351035
- [Background] Ferrara PE, Ronconi G, Viscito R, Pascuzzo R, Rosulescu E, Ljoka C, Maggi L, Ferriero G, Foti C. Efficacy of mesotherapy using drugs versus normal saline solution in chronic spinal pain: a retrospective study. Int J Rehabil Res. 2017 Jun;40(2):171-174. doi: 10.1097/MRR.0000000000000214. PMID 28125435
- [Background] Micarelli A, Viziano A, Augimeri I, Micarelli B, Capoccia D, Alessandrini M. Diagnostic route of cervicogenic dizziness: usefulness of posturography, objective and subjective testing implementation and their correlation. Disabil Rehabil. 2021 Jun;43(12):1730-1737. doi: 10.1080/09638288.2019.1680747. Epub 2019 Oct 26. PMID 31656108